CLINICAL TRIAL: NCT04364516
Title: Retrospective Observational Registry of Patients With Atrial Fibrillation From Vigo´s Health Area (Registro Observacional Retrospectivo de Pacientes Con Fibrilación Auricular Del Área de Vigo)
Brief Title: Retrospective Observational Registry of Patients With Atrial Fibrillation From Vigo´s Health Area
Acronym: CardioCHUVI-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Álvaro Cunqueiro (Other)
Responsible Party: Sponsor
Other Study IDs: HAC-ACO-2018-01
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrllation; Anticoagulation; Bleeding; Embolism.
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage; Embolism | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anticoagulation — Study of prognostic impact according to oral anticoagulation therapy (Vitamin K Antagonists or Direct Oral Anticoagulants)
  Other Names: Vitamin K Antagonists or Direct Oral Anticoagulants

SUMMARY:
Registry of all consecutive patients with atrial fibrillation from Heath Area of Vigo, since 2013 to 2020, in order to study therapy, mortality, cardiovascular complications and bleeding events.

DETAILED DESCRIPTION:
Retrospective observational registry of patients diagnosed of atrial fibrillation between 2013 and 2020. Clinical, analytical and echocardiographic data will be recorded, as well as therapeutic prescription information. Data on mortality and cardioembolic and hemorrhagic events will be collected during follow-up. The aim is to study the prevalence and incidence of atrial fibrillation, the anticoagulant treatment according to cardioembolic risk, the thromboembolic events and hemorrhagic events, the risk of mortality (Cardiovascular, Non-Cardiovascular), the contemporary management (Rhythm control versus frequency control strategy), and other complications, such as heart failure, acute coronary syndrome or cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed diagnoses of atrial fibrillation by ECG.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with atrial fibrillation from Health Area of Vigo
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2023-11-26 (Estimated)

PRIMARY OUTCOMES:
Mortality | Follow-up (3 years)
  All cause Mortality

SECONDARY OUTCOMES:
Bleeding | Follow-up (3 years)
  Bleeding according to International Society on Thrombosis and Haemostasis(ISTH) classiffication
Embolism | Follow-up (3 years)
  Embolic events include ischemic stroke, transient ischemic attack (TIA), pulmonary embolism (PE), and systemic embolism (SE). Ischemic stroke was defined as sudden onset of a focal deficit consistent with occlusion of a major cerebral artery (documented by means of magnet resonance imaging [MRI ]or computer tomography [CT]) and categorized. TIA was defined as a temporary neurologic deficit presumably due to reduced blood flow in a particular cerebral artery lasting for ≤24 hours with complete resolution of the neurologic deficit. A PE event was confirmed by spiral CT, perfusion-ventilation scan, pulmonary angiography, or autopsy) and resulted in a final PE diagnosis. A SE event was defined as any end-organ ischemia other than in the brain, heart, eyes, and lungs, caused by abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion in the absence of another likely mechanism.

CONTACTS AND LOCATIONS:
Overall Officials: EMAD ABU ASSI, PhD, MD, Study Director — University Hospital Alvaro Cunqueiro, Vigo, Spain; SERGIO RAPOSEIRAS ROUBIN, PhD, MD, Principal Investigator — University Hospital Alvaro Cunqueiro, Vigo, Spain; ANDRES IÑIGUEZ ROMO, PhD, MD, Study Chair — University Hospital Alvaro Cunqueiro, Vigo, Spain
Locations (1):
- Department of Cardiology, Hospital Álvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data of CardioCHUVI-AF registry could be merge with other registries, always they have similar characteristics, with a same registry nature

REFERENCES:
- [Derived] Abu-Assi E, Lizancos Castro A, Cespon-Fernandez M, Gonzalez-Bermudez I, Raposeiras Roubin S. Relative performance evaluation of four bleeding risk scores in atrial fibrillation patients. What does the new DOAC score provide? Int J Cardiol. 2024 Jul 15;407:132018. doi: 10.1016/j.ijcard.2024.132018. Epub 2024 Apr 3. PMID 38579940
- [Derived] Dominguez-Erquicia P, Raposeiras-Roubin S, Abu-Assi E, Bouzon-Iglesias P, Parada-Barcia JA, Lizancos-Castro A, Gonzalez-Garcia A, Noriega-Caro VA, Ledo-Pineiro A, Iglesias-Otero C, Gonzalez-Bermudez I, Iniguez-Romo A. Comparison of Outcomes in Patients With Atrial Fibrillation Under Oral Anticoagulation Therapy Analyzed by Body Weight (<60, 60 to 100, and >100 kg). Am J Cardiol. 2022 Dec 1;184:41-47. doi: 10.1016/j.amjcard.2022.07.028. Epub 2022 Sep 27. PMID 36175253
- [Derived] Raposeiras-Roubin S, Abu-Assi E, Lizancos Castro A, Barreiro Pardal C, Melendo Viu M, Cespon Fernandez M, Blanco Prieto S, Rossello X, Ibanez B, Filgueiras-Rama D, Iniguez Romo A. Nutrition status, obesity and outcomes in patients with atrial fibrillation. Rev Esp Cardiol (Engl Ed). 2022 Oct;75(10):825-832. doi: 10.1016/j.rec.2022.01.006. Epub 2022 Mar 9. English, Spanish. PMID 35279417
- [Derived] Cespon-Fernandez M, Raposeiras-Roubin S, Abu-Assi E, Melendo-Viu M, Garcia-Campo E, Iniguez-Romo A. Renin-Angiotensin System Inhibitors Prognostic Benefit in Older Patients with Atrial Fibrillation. J Am Med Dir Assoc. 2021 Oct;22(10):2190-2195. doi: 10.1016/j.jamda.2021.01.063. Epub 2021 Feb 16. PMID 33607060